CLINICAL TRIAL: NCT04526821
Title: Bovine Lactoferrin for the Prevention of COVID-19 Infection in Physicians and Nurses in Hospitals in Lima, Peru: a Double Blinded Randomized Clinical Trial (LF-COVID)
Brief Title: Lactoferrin for Prevention of COVID-19 in Health Care Workers
Acronym: LF-COVID
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was interrupted due to the arrival and distribution of the vaccine to hospital workers in Peru
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: Hospital Nacional Arzobispo Loayza (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SIDISI 202110
Record Dates: First submitted 2020-08-21; First posted 2020-08-26 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2020-08

CONDITIONS: SARS-CoV-2
Keywords: SARS-CoV-2 Infection; Lactoferrin; Health Care Workers
MeSH Terms: conditions — COVID-19 | interventions — Lactoferrin; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bovine Lactoferrin (Experimental): Bovine Lactoferrin plus standard measures of personal protection.
  Interventions: Drug: Bovine Lactoferrin
- Maltodextrin (Placebo Comparator): Maltodextrin plus standard measures of personal protection.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Drug: Bovine Lactoferrin — Bovine Lactoferrin 600mg daily for 12 weeks (3 chewable tablets of 100mg , twice a day), for 12 weeks plus personal portection provided from the hospital.
  Other Names: Lactoferrin
  Arms: Bovine Lactoferrin
Dietary Supplement: Maltodextrin — Maltodextrin 600mg daily for 12 weeks (3 chewable tablets of 100mg, twice a day), for 12 weeks plus personal portection provided from the hospital.
  Arms: Maltodextrin

SUMMARY:
Clinical trial in health care personnel (physicians, nurses or nurse assistants) to determine the effect of orally-administered bovine lactoferrin to prevent SARS-CoV-2 infection. Participants will be randomized to receive daily bovine lactoferrin plus standard measures during 12 weeks or placebo (maltodextrine) for the prevention of SARS-CoV-2. The target enrollment is 336 participants. Each study participant will be monitored twice a week for symptoms of COVID-19 and if symptoms occur, a RT-PCR will be performed. Additionally, we will evaluate asymptomatic infections, by measuring SARS-CoV-2 serology every 4 weeks.

DETAILED DESCRIPTION:
The SARS-CoV-2 infection has affected more than 100 countries around the world being classified as a pandemic by the World Health Organization. Health care providers are at high risk to become infected with the SARS-CoV-2 due to their continuous exposition to infected patients. Multiple strategies are being developed as potential prophylactic regimens, however to date (4th Aug 2020) none has proven to be effective for preventing the SARS-CoV-2 infection. Lactoferrin, an iron-binding protein with multiple physiological functions (anti-microbial, anti-inflammatory, and immunomodulatory), is one of the most important proteins present in mammalian milk. It has shown to inhibit the SARS entry to target cells by inhibiting the union of the SARS-CoV-2 spike protein with its receptor (ACE-II receptors), blocking the heparan sulfate proteoglycan receptor and it decreases the viral load of SARS-CoV-2 infecting culture cells in in vitro models. The study hypothesis is that lactoferrin given as a daily oral food supplement to health care workers will decrease the frequency of SARS-CoV-2 infection. The investigators will conduct a randomized double blinded placebo control clinical trial in physicians, nurses and nurse assistants who work in areas of care for patients with COVID-19 (emergency, hospitalization, and Intensive Care Unit) in hospitals in Lima, Peru, to determine the effect of bovine lactoferrin on the prevention of COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over 18 and under 60 years old
* Physicians or nurses or nurse assitant who work in areas of care for patients with COVID-19 (emergency, hospitalization, and Intensive Care Unit) in hospitals in Lima, Peru.
* Healthy participants, without COVID-19 suggestive symptoms
* Participant who wants to participate and signs the informed consent.

Exclusion Criteria:

* Participant who had a previous diagnosis of COVID-19.
* Participant positive in the initial screening for IgM or IgG or a positive RT-PCR for SARS-CoV-2.
* Participant with the following comorbidities: hypertension, coronary heart disease, diabetes mellitus, obesity, chronic lung disease, cancer, kidney failure, or other hematological disease.
* Pregnant woman.
* Participant that are part of another clinical trial or are taking any supplement or preventive treatment for COVID-19.
* Participant with known allergy to cow's milk protein.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 209 (Actual)
Dates: Start 2020-10-17 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Number of COVID-19 infections during the 12 weeks of intervention | Twelve weeks
  The primary study outcome will be defined by IgM, IgG and/or RT-PCR positivity for SARS-CoV 2.

SECONDARY OUTCOMES:
Severity of the COVID-19 infection | Twelve weeks
  Severity of SARS-CoV-2 infection (asymptomatic, mild, moderate, severe infection), assessed by the World Health Organization definitions
Duration of symptoms of the COVID-19 infection | Twelve weeks
  Duration of symptomatic SARS-CoV-2 infection defined by the number of days with SARS-CoV-2 symptomatology.
Frecuency of symptoms of the COVID-19 infection | Twelve weeks
  Frecuency of symptoms of SARS-CoV-2 infection: fever, fatigue, nonproductive cough, anorexia, myalgias, dyspnea, productive cough, taste and smell disorders, headache, rhinorrhea, nausea, diarrhea, and abdominal pain

CONTACTS AND LOCATIONS:
Overall Officials: Theresa J Ochoa, MD, PhD, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (2):
- Peru (2):
  - Hospital Nacional Arzobispo Loayza, Lima, Lim
  - Hospital Cayetano Heredia, Lima

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial, after deidentification, will be shared with researchers who provide a methodological sound study protocol previously approved by an independent ethics committee.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication of the study,
Access Criteria: Contact the study PI ( Theresa.ochoa@upch.pe)

REFERENCES:
- [Background] Legrand D. Overview of Lactoferrin as a Natural Immune Modulator. J Pediatr. 2016 Jun;173 Suppl:S10-5. doi: 10.1016/j.jpeds.2016.02.071. PMID 27234406
- [Background] Baker HM, Baker EN. A structural perspective on lactoferrin function. Biochem Cell Biol. 2012 Jun;90(3):320-8. doi: 10.1139/o11-071. Epub 2012 Jan 31. PMID 22292559
- [Background] Chang R, Ng TB, Sun WZ. Lactoferrin as potential preventative and adjunct treatment for COVID-19. Int J Antimicrob Agents. 2020 Sep;56(3):106118. doi: 10.1016/j.ijantimicag.2020.106118. Epub 2020 Jul 30. PMID 32738305
- [Background] Lang J, Yang N, Deng J, Liu K, Yang P, Zhang G, Jiang C. Inhibition of SARS pseudovirus cell entry by lactoferrin binding to heparan sulfate proteoglycans. PLoS One. 2011;6(8):e23710. doi: 10.1371/journal.pone.0023710. Epub 2011 Aug 22. PMID 21887302
- [Background] Campione E, Cosio T, Rosa L, Lanna C, Di Girolamo S, Gaziano R, Valenti P, Bianchi L. Lactoferrin as Protective Natural Barrier of Respiratory and Intestinal Mucosa against Coronavirus Infection and Inflammation. Int J Mol Sci. 2020 Jul 11;21(14):4903. doi: 10.3390/ijms21144903. PMID 32664543
- [Background] Mirabelli C, Wotring JW, Zhang CJ, McCarty SM, Fursmidt R, Frum T, Kadambi NS, Amin AT, O'Meara TR, Pretto CD, Spence JR, Huang J, Alysandratos KD, Kotton DN, Handelman SK, Wobus CE, Weatherwax KJ, Mashour GA, O'Meara MJ, Sexton JZ. Morphological Cell Profiling of SARS-CoV-2 Infection Identifies Drug Repurposing Candidates for COVID-19. bioRxiv [Preprint]. 2020 Dec 7:2020.05.27.117184. doi: 10.1101/2020.05.27.117184. PMID 32577649
- [Background] Marques de Carvalho CA, da Rocha Matos A, Caetano BC, de Sousa Junior IP, da Costa Campos SP, Geraldino BR, et al. In Vitro Inhibition of SARS-CoV-2 Infection by Bovine Lactoferrin [Internet]. Microbiology; 2020 May [cited 2020 May 25]. Available from: http://biorxiv.org/lookup/doi/10.1101/2020.05.13.093781
- [Derived] Navarro R, Paredes JL, Tucto L, Medina C, Angles-Yanqui E, Nario JC, Ruiz-Cabrejos J, Quintana JL, Turpo-Espinoza K, Mejia-Cordero F, Aphang-Lam M, Florez J, Carrasco-Escobar G, Ochoa TJ. Bovine lactoferrin for the prevention of COVID-19 infection in health care personnel: a double-blinded randomized clinical trial (LF-COVID). Biometals. 2023 Jun;36(3):463-472. doi: 10.1007/s10534-022-00477-3. Epub 2022 Dec 7. PMID 36474100